CLINICAL TRIAL: NCT00580099
Title: Assisted Exercise in Prematurity; Effects and Mechanisms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2005-4797; NIH Grant R01NR009070
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Growth; Development
Keywords: premature infant, body composition, total energy expenditure; inflammatory growth mediators
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 4 weeks of assisted exercise using passive range of motion on all major joints
  Interventions: Other: assisted exercise
- 2 (Active Comparator): cuddle for 20 minutes
  Interventions: Other: cuddle

INTERVENTIONS:
Other: assisted exercise — 4 weeks of passive range of motion exercise
  Arms: 1
Other: cuddle — cuddle infant for 20 minutes
  Arms: 2

SUMMARY:
Briefly our study is looking at the effects of 4 weeks of assisted exercise on the body composition and neurological/behavioral development of healthy growing premature infants enrolled between the ages of 30-33 weeks. It is a blinded study where the active group gets the exercise intervention and the control group is cuddled for the same amount of time -approximately 20 minutes. We get baseline data using muscle ultrasound, bone speed of sound and DEXA. We also get baseline blood samples to look at inflammatory mediators and growth hormone. Video of each subject is recorded an hour at two time points during the study to assess the babies for spontaneous activity. Nutritional intake information is collected daily and in the 4th week of the study assessments made for total energy expenditure using doubly labeled water. At this point in the study we repeat the ultrasounds and DEXA for comparison. Finally in the period just before discharge we do a complex neurological exam using the Brazelton NBAS assessment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at post menstrual ages of 23-33 weeks gestation Enrollment occurs at post menstrual age of 30 to 35 weeks.if their projected stay based on standard clinical criteria is four weeks after enrollment
* Enrollment occurs at post menstrual age of 30 up to 35 weeks, if their projected stay based on standard clinical criteria is 4 weeks after enrollment.
* Birth weight appropriate for gestational age (AGA) using current CDC growth charts. AGA is defined as plus or minus 2 standard deviations above the mean or above the third percentile.
* Tolerating full enteral feeds at greater than or equal to 100kcal/kg/day

Exclusion Criteria:

* Evidence of chromosomal or other major genetic abnormalities
* Existence of current diseases or syndromes including:

central nervous system or other neurological abnormalities chronic lung disease of prematurity requiring chronic use of corticosteroids, musculoskeletal diseases

* positive infant toxicology screen(urine) for drugs or alcohol
* Both parents are under the age of 18 years
* Babies with tracheostomy
* Babies receiving ventilator assistance with breathing
* Babies receiving IV fluids

Ages: 30 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Body composition, bone mineralization, muscle mass, anthropometric measurements | 4 weeks

SECONDARY OUTCOMES:
spontaneous movement | two time points
Neurological/behavioral status | end of 4th week
Blood Sampling to measure IGF-1, GHBP, IL-1ra | Baseline, week 2 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Dan M Cooper, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

REFERENCES:
- [Background] Gravem D, Lakes KD, Teran L, Rich J, Cooper D, Olshansky E. Maternal perceptions of infant exercise in the neonatal intensive care unit. J Obstet Gynecol Neonatal Nurs. 2009 Sep-Oct;38(5):527-33. doi: 10.1111/j.1552-6909.2009.01055.x. PMID 19883474
- [Result] Ahmad I, Zaldivar F, Iwanaga K, Koeppel R, Grochow D, Nemet D, Waffarn F, Eliakim A, Leu SY, Cooper DM. Inflammatory and growth mediators in growing preterm infants. J Pediatr Endocrinol Metab. 2007 Mar;20(3):387-96. doi: 10.1515/jpem.2007.20.3.387. PMID 17451077